CLINICAL TRIAL: NCT05157854
Title: Development and Process Evaluation of an Activity- and Recovery-oriented Intervention for People With Severe Mental Illness Living in Supported Housing - Active in My Home (AiMH)
Brief Title: Development and Evaluation of an Intervention (AiMH) for People With Severe Mental Illness Living in Supported Housing
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Active in My Home
Record Dates: First submitted 2021-11-15; First posted 2021-12-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Severe Mental Disorder
Keywords: Activity; Intervention; Occupational therapy; Severe mental illness; Supported accommodation; Recovery
MeSH Terms: conditions — Mental Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SH residents: Participants in the AiMH intervention
  Interventions: Behavioral: Active in My Home (AiMH)
- SH staff: Staff in the SH, acting as AiMH supporters

INTERVENTIONS:
Behavioral: Active in My Home (AiMH) — AiMH starts with two workshops for staff to introduce them to the intervention and the contributions expected from them. Their task is to participate in a couple of the sessions, inspire the course participant to stick to strategies developed during the sessions and support activity in general between the occupational therapy sessions.
  AiMH consists of eight sessions, five individual ones and three in a group. Each session has a theme, such as: "activity and health", and is built up with short lessons, using one's senses such as smell or touch, testing a simple activity, and setting goals for an activity one wants to test between sessions. The participants are given around 25 USD to try out that activity.
  Groups: SH residents

SUMMARY:
People with severe mental illness (SMI) spend a great amount of time in their homes. The home is thus of vital importance for an everyday life with meaningful activities. Systematic description of possibilities for meaningful activity in Supported Housing (SH) is however lacking. Even more importantly, support to meaningful activity in the SH context is sadly lacking. That there is a need for support to activity for those who live in SH is partly evident from research, but has also become obvious through several contacts between the investigators' research group and staff working in SH settings.

In a first step the investigators described how people with SMI use their time while being at home and how the participants perceive their possibilities for being active. Comparisons were made with people with SMI who had ordinary housing and got housing support. A mixed-methods approach with well-established rating scales and qualitative interviews was used.

The current study aims are to:

1. Based on the findings from Step 1 above, develop an intervention for those who live in SH. The intervention goal is to increase the possibilities for satisfying engagement in activities in one's home. The intervention will also build on previous experiences form developing and evaluating interventions for the target group.
2. Investigate what changes people who participate in such an intervention will make regarding engagement in activities, satisfaction with activities, recovery from mental illness, self-rated health, and quality of life.
3. Investigate how users and staff perceive the SH services' possibilities to offer or stimulate to different types of activity, as well as their satisfaction with the new intervention.

People with SMI are a sadly neglected group with respect to access to meaningful activities. Enriching supported with features that enable more meaningful activity in the home context could lead to gains for the individual (increased well-being) as well as society (better services and decreased needs for support). The project is of relevance for both persons with SMI and society through its emphasis on 1) well-being among people with substantial functional limitations and 2) a meaningful everyday life in the intersection between housing and activity.

DETAILED DESCRIPTION:
Background and Main Purpose People with severe mental illness (SMI) say that being active and taking part in social interaction are the most essential elements for being able to experience meaning in life. Interventions and research into activity for this target group have so far been concentrated on work rehabilitation and on meaningful activities in community-based activity centres. The common denominator here is the assumption that the individual leaves their residence in order to engage in activities. The focus of this application is, however, on the individual's situation in their home environment. The latter can vary from living in one's own apartment/ house without support, often termed ordinary housing, to supported housing (SH), which links housing and support and is situated in supervised group homes or apartments located in one building. An intermediate form is housing support, which is when a person living in an ordinary home receives support in order to manage that situation.

The home is of fundamental importance for the possibilities for people with SMI to lead an everyday life characterized by meaningful activities, being as this group spend a greater part of their time in the home setting. Activity in one's home is also linked with occupational engagement in other social and geographical contexts. There is a lack of interventions aiming at improving the possibilities for an active and engaged everyday life within the frame of the home setting and the near neighbourhood. The need for support in this field is evident from the research literature, but has also emerged in countless contacts between the investigator's research group and staff working with supported housing and housing support for people with SMI.

The current project is Step two of research aiming to promote meaningful and engaging activities in the home setting for people with SMI in SH, and thereby also support their health, well-being and recovery. Step 1 was a survey of how people with SMI who live in SH, compared to those who receive housing support in an ordinary home, used their time while in their homes and how the participants experienced their opportunities for activity. Findings revealed that the residents had a low activity level and were often alone. The conclusion was that services need to support individually adjusted contextual stimuli and individualize the support to help residents find a good balance and motivate them to be active in and outside SH, which can support a recovery process. Against this background, the aims of Step 2 are to:

* Design an intervention for those who live in SH, on the basis of Step 1 and previous research on activity- and recovery-based interventions, for increasing the residents' opportunities for satisfactory engagement in everyday activities.
* Evaluate the intervention by mixed methods, including an uncontrolled quantitative study and qualitative studies.

Survey of the field Research on SH and housing support for people with SMI has developed during the last years. The focus has been on comparing institutional and community living and on the individual's preferences as to how SH residents wish to live. The participants' views on their living arrangements and on aspects of the physical and psychosocial environments have also been examined. However, research on activities in the home environment has received very little attention in Sweden and internationally, although Priebe et al. reported on how support from the staff was adjusted to promote self-care activities in SH in Great Britain. A small-scale study in Sweden found that rehabilitation, which was based on occupational therapy and client-centeredness and aimed at increased activity in the SH context, resulted in good progress regarding both activity and health-related factors. The improvements were seen to be maintained in a six-month follow-up perspective thus indicating that this was a promising intervention. Only 17 participants were included in that study, however, which makes generalisation impossible.

Activity is defined, in the present application, as everyday life activities in a broad sense, including work-related activities, household work, self-care, and all kinds of recreational activities (physical, cultural and social). Whereas work-related activities are mainly performed outside the home, taking care of one's home, self-care and leisure activities often take place in the home. There is convincing evidence of a strong connection between on the one hand satisfying and engaging activities, and on the other health and well-being. This makes it important to find the best support for meaningful activities and engaging activities in different areas of life, in the home as well as in activity centres and in relation to working life.

Previous research indicates that the residents in SH are those who have the most severe SMI and the activity level in that context is very low. Bejerholm and Eklund found that people with schizophrenia, some of whom lived in SH, spent a great deal of time at home, alone, and with a very limited repertoire of activities, very often spending time lying resting and thinking, watching TV, and smoking. Those living in ordinary housing were engaged in public activities to a greater extent than those receiving different kinds of housing services. It also appeared that those who were more strongly engaged in activities were more satisfied with current housing conditions and level of independence. Research has also shown that housing with optimal support can promote recovery from mental illness. Based on the above and since meaningful activity is an important aspect of recovery from mental illness, it is obvious that further descriptive and comparative research is important for identifying subgroups and activity areas where support is needed to enable meaningful, engaging and satisfactory activities in the home setting and the near environment.

Residents in SH are a vulnerable group with a great need for support. The fact that people with SMI often lead isolated and passive lives makes it important to consider efforts that can support a more meaningful life for SH residents. Such efforts can also include staff to accomplish the best possible impact. Research has shown that preconceptions about support and activity among staff working in SH are of importance for how the support measures are designed in practice.

Study Design

The current project will answering the following research questions:

1. Considering the results from Step 1 and previous experience from evaluating interventions for the target group, what are the implications for the development of an intervention, within the context of SH, in order to improve the opportunities for creating a satisfying engagement in everyday activities? How can such an intervention be designed?
2. What changes will people who participate in such an intervention make regarding engagement in activities, satisfaction with activities, recovery from mental illness, self-rated health, and quality of life?
3. How do users and staff perceive the housing services' possibilities to offer or stimulate to different types of activity, and what is their satisfaction with the new intervention? From now on, that intervention is termed Active in my Home (AiMH).

Methods The project will be based on mixed methods and be using both quantitative and qualitative methodology. Trained research assistants will perform the data collection.

No precisely comparable study can be used as a basis for the power calculation, but we consider the SDO instrument, which assesses satisfaction with everyday occupations, to be an adequate measure for a power analysis. A study found a mean difference of 0.5 points on the SDO between groups of people with mental illness who had varying structure to their everyday life. Based on the means and standard deviations from that study, we recently made power calculations for another study and arrived at 41 participants in each group as the desired sample size to detect a difference on the SDO of 0.5 with 80% power at p<0.05. Since that study seemed somewhat underpowered we aim to include 60 residents. The number of staff will be what is available; we invite those who work with the 60 residents who have agreed to participate in the AiMH intervention.

The participants will be investigated with well tested instruments with good psychometric qualities.

In addition, qualitative studies will be made in order to gain a greater understanding of the possibilities of providing meaningful and engaging activities in the home context. Focus groups with users are planned in order to stimulate reflection and discussion. The transcripts will be analysed by latent content analysis.

The uncontrolled evaluation (questions b and c above) will include three measurement points: a baseline before the intervention, post-measurement after competed intervention and follow-up measurement 6-9 months later. SH units will be sought in various geographical areas in southern, western and eastern Sweden. Residents who meet the criteria of: having a severe mental illness (> 2 years of contact with psychiatric services and an estimated level of functioning of < 50 on the GAF scale), not having substance abuse as the main diagnosis, not having comorbidity of dementia or intellectual disability, and being able to speak and understand Swedish will be invited. SH units in the public sector as well as the private sector will be invited. We plan to include 10 units to start with. The inclusion of new SH units will go on until the desired sample of 60 participants has been obtained. By inviting staff who support these participants, we estimate that about the same number of staff members (=60) will be enrolled.

Qualitative interviews will be performed to gain a deeper insight into the perceptions of the AIMH intervention of the residents, the staff and the significant others. Not to intervene with the AIMH intervention, the interviews (audiotaped) will be made after completed follow-ups. The idea is to perform individual interviews to catch residents' experiences, but focus groups with staff to stimulate reflection and discussion. The interview data will be transcribed and analyzed with qualitative content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Residents: having a severe mental illness (> 2 years of contact with psychiatric services and an estimated level of functioning of < 50 on the GAF scale); good command of the Swedish language
* Staff: supporting one or more residents who take part in the AiMH intervention

Exclusion Criteria:

* Residents: having substance abuse as the main diagnosis; comorbidity of dementia or intellectual disability,

Staff: Not having had any contact with AiMH participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SH units will be sought in various geographical areas in southern, western and eastern Sweden. Residents who meet the criteria of:will be invited. We plan to include 10 units to start with and go on until the desired sample of 60 participants has been obtained. By inviting staff who support these participants, we estimate that about the same number of staff members (=60) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Profiles of Occupational Engagement in people with Severe Mental Illness (POES) Profiles of Occupational Engagement in people with Severe Mental Illness | At baseline
  Interview-based time-use diary covering the past 24 hours. The diary sheet has five columns, one for each of: 1) time slot, 2) type of activity, 3) where the activity is performed, 4) with whom, and 5) any feelings or reflections.
Profiles of Occupational Engagement in people with Severe Mental Illness (POES) Profiles of Occupational Engagement in people with Severe Mental Illness | After 12 weeks of AiMH intervention
  Interview-based time-use diary covering the past 24 hours. The diary sheet has five columns, one for each of: 1) time slot, 2) type of activity, 3) where the activity is performed, 4) with whom, and 5) any feelings or reflections.
Profiles of Occupational Engagement in people with Severe Mental Illness (POES) Profiles of Occupational Engagement in people with Severe Mental Illness | At a 6 - 9 month follow-up
  Interview-based time-use diary covering the past 24 hours. The diary sheet has five columns, one for each of: 1) time slot, 2) type of activity, 3) where the activity is performed, 4) with whom, and 5) any feelings or reflections.
Questionnaire about Personal Recovery (QPR) Profiles of Occupational Engagement in people with Severe Mental Illness | At baseline
  The individual's evaluation of his/her recovery from mental illness. A higher score means a better outcome
Questionnaire about Personal Recovery (QPR) Profiles of Occupational Engagement in people with Severe Mental Illness | After 12 weeks of AiMH intervention
  The individual's evaluation of his/her recovery from mental illness. A higher score means a better outcome.
Questionnaire about Personal Recovery (QPR) Profiles of Occupational Engagement in people with Severe Mental Illness | At a 6 - 9 month follow-up
  The individual's evaluation of his/her recovery from mental illness. A higher score means a better outcome.

SECONDARY OUTCOMES:
Brief Inspire | At baseline + after 12 weeks of AiMH intervention + at a 6 - 9 month follow-up.
  Questionnaire reflecting perceived support from the mental health worker. A higher score means a better outcome.
Satisfaction with AiMH | After 12 weeks of AiMH intervention.
  Questionnaire reflecting Satisfaction with AiMH. A higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Bejerholm, PhD, Study Director — Lund University, Dept of Health Sciences

IPD SHARING:
Plan to Share IPD: No
According to Swedish law, "Act (2003:460) concerning the Ethical Review of Research Involving Humans", data must not be shared outside of the research team. In publications we will state that data can be shared on reasonable request.

REFERENCES:
- [Background] Tjornstrand C, Eklund M, Bejerholm U, Argentzell E, Brunt D. A day in the life of people with severe mental illness living in supported housing. BMC Psychiatry. 2020 Oct 15;20(1):508. doi: 10.1186/s12888-020-02896-3. PMID 33059664
- [Background] Eklund M, Argentzell E, Bejerholm U, Tjornstrand C, Brunt D. Wellbeing, activity and housing satisfaction - comparing residents with psychiatric disabilities in supported housing and ordinary housing with support. BMC Psychiatry. 2017 Aug 30;17(1):315. doi: 10.1186/s12888-017-1472-2. PMID 28854907
- [Derived] Eklund M, Tjornstrand C. Resident and staff perceptions of an activity- and recovery-based intervention in supported housing for people with severe mental illness - a longitudinal pilot study. BMC Psychiatry. 2022 Jun 16;22(1):404. doi: 10.1186/s12888-022-04050-7. PMID 35710347